CLINICAL TRIAL: NCT07115641
Title: A Multicenter Clinical Randomized Controlled Trial on the Efficacy and Safety of Huoluo Pills Combined With Iguratimod Tablets in the Treatment of Rheumatoid Arthritis
Brief Title: Clinical Trial of Huoluo Pills Combined With Iguratimod Tablets in the Treatment of Rheumatoid Arthritis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wangjing Hospital, China Academy of Chinese Medical Sciences (Other)
Collaborators: Institute of Science, Beijing Tongrentang Co., Ltd. (Unknown); Beijing Leadingpharm Medicine Technology Development (Unknown); Shanghai Guanghua Hospital of Integrated Traditional Chinese and Western Medicine (Other); The Second Affiliated Hospital of Guizhou University of Traditional Chinese Medicine (Unknown); The First Affiliated Hospital of Henan university of CM (Unknown); Xi'an No.5 Hospital (Unknown); Liaoning University of Traditional Chinese Medicine Affiliated Hospital (Unknown); Affiliated Hospital of Shandong University of Traditional Chinese Medicine (Other); Affiliated Hospital of Shanxi University of Chinese Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: leadingpharm2025002; ITMCTR2025000953 (Other: ITMCTR); MR-11-25-036909 (Other: China National Medical Research Registration and Filing Information System)
Record Dates: First submitted 2025-07-21; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-06

CONDITIONS: Rheumatoid Arthritis
Keywords: Huoluo Pills; Iguratimod Tablets
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — iguratimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trial group (Experimental): Huoluo Pills + Iguratimod Tablets
  Interventions: Drug: Huoluo Pills; Drug: Iguratimod Tablets
- Control group (Other): Iguratimod Tablets
  Interventions: Drug: Iguratimod Tablets

INTERVENTIONS:
Drug: Huoluo Pills — Huoluo Pills: Orally take 1 pill once, twice a day (swallow with warm water)
  Arms: Trial group
Drug: Iguratimod Tablets — Iguratimod Tablets: Orally take 1 tablet once, twice a day (one tablet in the morning and one in the evening, after meals)

SUMMARY:
This study aims to systematically evaluate the efficacy and safety of Huoluo Pills combined with Iguratimod Tablets in the treatment of rheumatoid arthritis (RA). A total of 240 patients with RA belonging to the syndromes of Wind - Damp Obstruction or Cold - Damp Obstruction will be enrolled in 8 centers (randomly assigned to groups). The experimental group will receive oral Huoluo Pills combined with Iguratimod Tablets, while the control group will receive oral Iguratimod Tablets alone. Both groups will be administered continuously for 12 weeks.

Primary Efficacy Index: The proportion of ACR20 responders in each group at the end of treatment.

Key Secondary Efficacy Index: The change in DAS28 (CRP) score from baseline in each group at the end of treatment.

Other Secondary Efficacy Indexes: RF, CRP, ESR, IL - 6, ACR50, ACR70, CDAI, SDAI, HAQ - DI, SF - 36, FACIT - Fatigue, and Traditional Chinese Medicine (TCM) syndrome scores.

Safety Indexes: Physical examination, blood routine, urine routine, blood biochemistry, coagulation function, etc.

This study will investigate the efficacy and safety of Huoluo Pills combined with Iguratimod Tablets in the treatment of RA with Wind - Damp Obstruction or Cold - Damp Obstruction syndromes.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who meet the Western medicine classification criteria for rheumatoid arthritis (RA) launched by the American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) in 2010 and have been clearly diagnosed with RA.
2. Subjects who meet the diagnostic criteria for traditional Chinese medicine syndromes of "Wind-Dampness Obstruction Syndrome (Main symptoms: ① Joint pain and swelling wandering; ② Joint pain and swelling intermittent. Secondary symptoms: ① Aversion to wind or sweating; ② Headache; ③ Heaviness of the limbs. Tongue and pulse manifestations: Pale red tongue thin white coating slippery or floating pulse. Diagnosis can be made by having 2 main symptoms or 1 main symptom + 2 secondary symptoms combined with the tongue and pulse manifestations)" or "Cold-Dampness Obstruction Syndrome (Main symptoms: ① Cold joint pain the joints feel cold to the touch and the skin color is not red; ② The pain worsens when exposed to cold and alleviates when warmed. Secondary symptoms: ① Joint stiffness limited flexion and extension; ② Cold limbs or aversion to cold and preference for warmth; ③ Bland taste in the mouth without thirst. Tongue and pulse manifestations: Enlarged tongue body pale tongue white or greasy coating wiry or tight pulse. Diagnosis can be made by having 2 main symptoms or 1 main symptom + 2 secondary symptoms combined with the tongue and pulse manifestations)".
3. Subjects with a Disease Activity Score in 28 joints (DAS28) (ESR) score > 2.6 and ≤ 5.1 or a DAS28 (CRP) score > 2.3 and ≤ 4.1.
4. Male or female subjects aged ≥ 18 years old and ≤ 70 years old.
5. Subjects who have not used iguratimod and Huoluo Pills within 4 weeks before the first administration of the investigational drug.
6. If the subject is receiving treatment with traditional disease-modifying antirheumatic drugs (DMARDs) during screening monotherapy with one of methotrexate (MTX) leflunomide or hydroxychloroquine is allowed and the dosage should be stable for at least 12 weeks before the first administration of the investigational drug (MTX dosage ≤ 15 mg/week leflunomide ≤ 20 mg/day hydroxychloroquine ≤ 400 mg/day).
7. Subjects who are receiving treatment with non-steroidal anti-inflammatory drugs (NSAIDs) during screening should have a stable dosage for at least 2 weeks before the first administration of the investigational drug and maintain the same dosage during the trial.
8. Subjects who are receiving hormone treatment during screening should have a stable condition (limited to oral administration of ≤ 10 mg/d prednisone acetate or equivalent dose) for at least 4 weeks before the first administration of the investigational drug and maintain stable treatment during the trial.
9. Subjects who voluntarily agree to participate in this trial sign a written informed consent form are able to follow the visit and related procedures specified in the protocol and have good compliance.

Exclusion Criteria:

1. Those who have used plant medicine preparations such as Tripterygium glycosides total glucosides of paeony sinomenine or other traditional Chinese medicine preparations that affect the evaluation of the therapeutic effect within 4 weeks before the first administration of the test drug;
2. Those who have received intramuscular injection intravenous injection or intra-articular injection of glucocorticoid treatment within 4 weeks before the first administration of the test drug;
3. Patients who have received treatment with biological agents within 12 weeks before the first administration of the test drug;
4. Those who suffer from active gastrointestinal diseases (such as peptic ulcers) severe interstitial lung diseases low bone marrow function severe cardiovascular and cerebrovascular diseases (such as acute myocardial infarction unstable angina pectoris intracerebral hemorrhage transient ischemic attack) severe organic lesions such as poorly controlled diabetes mellitus or those who have a history of malignant tumors in the past 5 years or those with mental illnesses. ;
5. Those known to have tuberculosis HIV hepatitis B hepatitis C syphilis or other active or chronic persistent infections;
6. Those who are allergic to the drugs involved in the research protocol or have contraindications to their use;
7. Those who have received live vaccines within 4 weeks before screening or inactivated vaccines within 2 weeks before screening or those who have a vaccination plan during the trial;
8. Those with any of the following conditions in the auxiliary examination during screening: 1) AST or ALT > 1.5 times the upper limit of the normal reference value or the estimated glomerular filtration rate (eGFR) ≤ 60 mL/min/1.73m²; 2) Hemoglobin < 90 g/L or white blood cell count < 3.0×10⁹/L or neutrophil count < 1.5×10⁹/L or lymphocyte count < 0.5×10⁹/L or platelet count < 90×10⁹/L;
9. Pregnant or lactating women those with a fertility plan or those planning to donate sperm or eggs;
10. Those who are participating in other clinical trials before screening;
11. Those whom the investigator deems to have other factors that make them unsuitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-08-11 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of subjects achieving ACR20 | At the end of the treatment (on the 84th day)
  ACR20: The improvement degree of the number of tender joints and the number of swollen joints is ≥20%, and the improvement degree of at least 3 items among the remaining 5 items is ≥20%.

SECONDARY OUTCOMES:
The change of Disease Activity Score in 28 Joints-C-Reactive Protein（DAS28-CRP） score compared with the baseline | At the end of the treatment (on the 84th day)
  DAS28-CRP=0.56×sqrt（TJC28）+0.28×sqrt（SJC28）+0.36×ln（CRP+1）+0.014×GH+0.96
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * ESR: Erythrocyte Sedimentation Rate;
  * CRP: C-reactive Protein;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity DAS28-CRP thresholds:
  * High: > 4.1;
  * Moderate: > 2.7 and ≤ 4.1;
  * Low: > 2.3 and ≤ 2.7;
  * Remission: ≤ 2.3
The proportion of subjects achieving ACR20 | By the 28th day of treatment
  ACR20: The improvement degree of the number of tender joints and the number of swollen joints is ≥20%, and the improvement degree of at least 3 items among the remaining 5 items is ≥20%.
The change of Disease Activity Score in 28 Joints-C-Reactive Protein（DAS28-CRP） score compared with the baseline | By the 28th day of treatment
  DAS28-CRP=0.56×sqrt（TJC28）+0.28×sqrt（SJC28）+0.36×ln（CRP+1）+0.014×GH+0.96 - TJC28: Number of tender joints among 28 joints; - SJC28: Number of swollen joints among 28 joints; - ESR: Erythrocyte Sedimentation Rate; - CRP: C-reactive Protein; - GH: Patient's global assessment of disease activity (VAS score, unit: 100mm). Disease activity DAS28-CRP thresholds: - High: > 4.1; - Moderate: > 2.7 and ≤ 4.1; - Low: > 2.3 and ≤ 2.7; - Remission: ≤ 2.3
The remission rate of Disease Activity Score in 28 Joints-C-Reactive Protein（DAS28-CRP） | When treating up to the 28th and 84th days
The low activity rate of Disease Activity Score in 28 Joints-C-Reactive Protein（DAS28-CRP） | When treating up to the 28th and 84th days
The remission rate of Disease Activity Score in 28 Joints-Erythrocyte Sedimentation Rate（DAS28-ESR） | When treating up to the 28th and 84th days
The low activity rate of Disease Activity Score in 28 Joints-Erythrocyte Sedimentation Rate（DAS28-ESR） | When treating up to the 28th and 84th days
The change of Disease Activity Score in 28 Joints-Erythrocyte Sedimentation Rate（DAS28-ESR） score compared with the baseline | When treating up to the 28th and 84th days
  DAS28-ESR=0.56×sqrt（TJC28）+0.28×sqrt（SJC28）+0.70×ln（ESR）+0.014×GH
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * ESR: Erythrocyte Sedimentation Rate;
  * CRP: C-reactive Protein;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity DAS28-ESR thresholds:
  * High: > 5.1;
  * Moderate: > 3.2 and ≤ 5.1;
  * Low: > 2.6 and ≤ 3.2;
  * Remission: ≤ 2.6
The proportion of subjects with ACR50 | When treating up to the 28th and 84th days
  ACR50: The improvement degree of the number of tender joints and the number of swollen joints is ≥50%, and the improvement degree of at least 3 items among the remaining 5 items is ≥50%.
The proportion of subjects with ACR70 | When treating up to the 28th and 84th days
  ACR70: The improvement degree of the number of tender joints and the number of swollen joints is ≥70%, and the improvement degree of at least 3 items among the remaining 5 items is ≥70%.
The proportion of subjects with a CDAI（Clinical Disease Activity Index） score ≤ 10 | When treating up to the 28th and 84th days
  CDAI=（TJC28+SJC28+GH+EH）/4
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm);
  * EH: Physician's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity thresholds:
  * High: > 22;
  * Moderate: > 10 and ≤ 22;
  * Low: > 2.8 and ≤ 10;
  * Remission: ≤ 2.8.
The proportion of subjects with a CDAI（Clinical Disease Activity Index） score ≤ 2.8 | When treating up to the 28th and 84th days
  CDAI=（TJC28+SJC28+GH+EH）/4 - TJC28: Number of tender joints among 28 joints; - SJC28: Number of swollen joints among 28 joints; - GH: Patient's global assessment of disease activity (VAS score, unit: 100mm); - EH: Physician's global assessment of disease activity (VAS score, unit: 100mm). Disease activity thresholds: - High: > 22; - Moderate: > 10 and ≤ 22; - Low: > 2.8 and ≤ 10; - Remission: ≤ 2.8.
The change of CDAI（Clinical Disease Activity Index） score compared with the baseline | When treating up to the 28th and 84th days
  CDAI=（TJC28+SJC28+GH+EH）/4 - TJC28: Number of tender joints among 28 joints; - SJC28: Number of swollen joints among 28 joints; - GH: Patient's global assessment of disease activity (VAS score, unit: 100mm); - EH: Physician's global assessment of disease activity (VAS score, unit: 100mm). Disease activity thresholds: - High: > 22; - Moderate: > 10 and ≤ 22; - Low: > 2.8 and ≤ 10; - Remission: ≤ 2.8.
The proportion of subjects with an SDAI（Simplified Disease Activity Index） score ≤ 11 | When treating up to the 28th and 84th days
  SDAI=（TJC28+SJC28+CRP+GH+EH）/5
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * CRP: C-reactive Protein;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm);
  * EH: Physician's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity thresholds:
  * High: > 26;
  * Moderate: > 11 and ≤ 26;
  * Low: > 3.3 and ≤ 11;
  * Remission: ≤ 3.3.
The proportion of subjects with an SDAI （Simplified Disease Activity Index）score ≤ 3.3 | When treating up to the 28th and 84th days
  SDAI=（TJC28+SJC28+CRP+GH+EH）/5
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * CRP: C-reactive Protein;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm);
  * EH: Physician's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity thresholds:
  * High: > 26;
  * Moderate: > 11 and ≤ 26;
  * Low: > 3.3 and ≤ 11;
  * Remission: ≤ 3.3.
Change in SDAI （Simplified Disease Activity Index）score from baseline | When treating up to the 28th and 84th days
  SDAI=（TJC28+SJC28+CRP+GH+EH）/5
  * TJC28: Number of tender joints among 28 joints;
  * SJC28: Number of swollen joints among 28 joints;
  * CRP: C-reactive Protein;
  * GH: Patient's global assessment of disease activity (VAS score, unit: 100mm);
  * EH: Physician's global assessment of disease activity (VAS score, unit: 100mm).
  Disease activity thresholds:
  * High: > 26;
  * Moderate: > 11 and ≤ 26;
  * Low: > 3.3 and ≤ 11;
  * Remission: ≤ 3.3.
The change of HAQ-DI（Health Assessment Questionnaire-Disability Index Score） score compared with the baseline | When treating up to the 28th and 84th days
  The HAQ-DI scale consists of 20 questions, each scored on a 4-point scale: 0 points for "no difficulty", 1 point for "some difficulty", 2 points for "great difficulty", and 3 points for "unable to perform". The total score is 0-60 points.The higher the score, the worse the function or mood.
The changes of the scores of each dimension of the quality of life (SF-36,36-item Short-Form) compared with the baseline respectively. | When treating up to the 28th and 84th days
  1. Calculation of raw scores:
     For each question, assign the corresponding score according to the answer option. Usually, the options are arranged in the order from "best" to "worst" and given corresponding score values (such as a 5-point scale, 4-point scale, or 3-point scale).
     Calculate the total raw score for each dimension.
  2. Calculation of converted scores:
  Since the number of questions and score ranges in different dimensions may vary, it is necessary to convert raw scores into standard scores (i.e., converted scores) for comparison and analysis.
  The calculation method of converted scores is usually: (Raw score - Minimum possible raw score of the dimension) / (Maximum possible raw score of the dimension - Minimum possible raw score of the dimension) × 100.
  In this way, the converted score of each dimension will be standardized between 0 and 100, facilitating comparison and analysis.
  A higher score indicates a better state of health.
The change of the Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) score in disease treatment compared with the baseline. | When treating up to the 28th and 84th days
  The FACIT-Fatigue consists of 13 questions, each scored on a 5-point scale (0-4 points), with a total score ranging from 0 to 52 points. A higher score indicates a more severe degree of fatigue in the patient.
The change of TCM syndrome score compared with the baseline and the effective rate | When treating up to the 28th and 84th days
  The scale scores corresponding to the primary symptoms are 0, 2, 4, and 6 points respectively, and the scale scores corresponding to the secondary symptoms are 0, 1, 2, and 3 points respectively. A higher score indicates more obvious symptoms.
  Criteria for Therapeutic Effect of TCM Syndromes:
  1. Clinical cure: TCM-related syndromes disappear or basically disappear, and the reduction of syndrome scores is ≥95%;
  2. Marked effect: TCM-related syndromes are significantly improved, with a reduction of syndrome scores >95% and ≥70%;
  3. Effective: TCM-related syndromes are improved, with a reduction of syndrome scores >70% and ≥30%;
  4. Ineffective: TCM-related syndromes show no significant improvement or even worsen, with a reduction of syndrome scores <30%.
  Total effective rate = [(Number of cured cases + Number of markedly effective cases + Number of effective cases) / Total number of cases] × 100%
The change of the Visual Analogue Scale (VAS) score of the doctor's overall assessment of disease activity (EH) compared with the baseline. | When treating up to the 28th and 84th days
  The VAS score ranges from 0 to 100 mm, where 0 represents no pain or no activity, and 100 represents the most severe.
The change of the Visual Analogue Scale (VAS) score of the subjects' assessment of articular pain (PtAAP) compared with the baseline. | When treating up to the 28th and 84th days
  The VAS score ranges from 0 to 100 mm, where 0 represents no pain or no activity, and 100 represents the most severe.
The change of the Visual Analogue Scale (VAS) score of the subjects' overall assessment of disease activity (GH) compared with the baseline. | When treating up to the 28th and 84th days
  The VAS score ranges from 0 to 100 mm, where 0 represents no pain or no activity, and 100 represents the most severe.
The change of the detected value of C-reactive protein (CRP) compared with the baseline. | When treating up to the 28th and 84th days
The change of the detected value of erythrocyte sedimentation rate (ESR) compared with the baseline | When treating up to the 28th and 84th days
The change of rheumatoid factor (RF) compared with the baseline | By the 84th day of treatment
The change of the inflammatory factor interleukin - 6 (IL - 6) compared with the baseline. | By the 84th day of treatment
The changes of coagulation - related indexes compared with the baseline. | By the 84th day of treatment
The dosage of Loxoprofen Sodium Tablets | When treating up to the 28th and 84th days

IPD SHARING:
Plan to Share IPD: No